CLINICAL TRIAL: NCT02007057
Title: Prospective Randomized Comparative Study of the Effectiveness of Suprascapular Nerve Block in Arthroscopic Shoulder Surgery
Brief Title: Effectiveness of Suprascapular Nerve Block in Arthroscopic Shoulder Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Ambroise Paré Paris (Other)
Responsible Party: Principal Investigator, Shahnaz Klouche, MD, Physician Responsible of Clinical Research, Hospital Ambroise Paré Paris
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APR112013
Record Dates: First submitted 2013-11-29; First posted 2013-12-10 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Rotator Cuff Tear; Pain
Keywords: Suprascapular nerve block; Interscalene nerve block
MeSH Terms: conditions — Rotator Cuff Injuries; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interscalene nerve block (Active Comparator): Interscalene block is performed preoperatively with ultrasound guidance and neurostimulation 0.8 milliampere. The block is performed using "in-plane" approach with a needle of 50 mm for a neurostimulation. During the injection, it is verified that the diffusion extends to the anterior and posterior space. If the posterior distribution is limited, the needle is remobilized to obtain an overall diffusion: a bolus of 20 mL of ropivacaine 0.75% is made by the anesthetist. The effectiveness of the nerve block is checked before the start of surgery.
  Interventions: Procedure: Interscalene nerve block
- Suprascapular nerve block (Experimental): The suprascapular block is performed at the end of surgery when the incisions are closed but before the removal of the surgical drapes. The material used is a compound of a 10 cc syringe sterile equipment, a green intramuscular needle (14 gauge) and a bulb 10 cc of 0.75% Ropivacaine. The injection of 10 cc is realized by the technical princeps
  Interventions: Procedure: Suprascapular nerve block

INTERVENTIONS:
Procedure: Suprascapular nerve block
  Arms: Suprascapular nerve block
Procedure: Interscalene nerve block
  Arms: Interscalene nerve block

SUMMARY:
Most arthroscopic surgeries of the shoulder are currently performed as an outpatient. The postoperative analgesia should be optimal. General anesthesia allows for any arthroscopic surgery but does not provide a satisfactory postoperative analgesia . The locoregional anesthesia is recommended and includes several techniques: the interscalene nerve block, the suprascapular nerve block, intra-articular injection of local anesthetic and subacromial infiltration. The interscalene nerve block is currently the gold standard for anesthesia and postoperative analgesia for arthroscopic shoulder surgery with a success rate above 80% . However it must be carried out by teams experienced in the locoregional anesthesia because it is operator -dependent. The suprascapular nerve block is a simple technique that can be performed by the surgeon after surgery , effective in arthroscopic shoulder surgery , less invasive than the interscalene nerve block and exposing the patient to fewer complications. However, his interest was not assessed in the repair of tendons of the rotator cuff. The main hypothesis of this study is that the suprascapular nerve block is as effective as the interscalene nerve block in the prevention of early postoperative pain after arthroscopic repair of the infra and / or the supraspinatus rotator cuff tendons, without increasing the analgesic consumption while reducing the risk of complications related to regional anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years
* Arthroscopic repair of infra and / or supraspinatus tendon of the rotator cuff with or without associated procedure on the biceps, the acromion-clavicular joint or acromion
* Informed consent

Exclusion Criteria:

* Allergy to local anesthetics (ropivacaine, bupivacaine, xylocaine)
* Previous surgery on the involved shoulder
* Severe or morbid obesity (BMI> 35)
* Psychiatric disorders (impossible self-assessment of the pain)
* Patient unfit physically, mentally or legally to give informed consent
* Patient refusal
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Self-assessment of the mean shoulder pain | Visual analog scale (VAS) during 2 days postoperatively

SECONDARY OUTCOMES:
Self assessment of shoulder pain | VAS twice daily during the first postoperative week
Complications of locoregional anesthesia | Yes or No during the first 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Hardy, MD, PhD, Principal Investigator — Ambroise Pare Hospital
Locations (1):
- Hopital Ambroise Pare, Boulogne-Billancourt, France